CLINICAL TRIAL: NCT00006034
Title: A Randomized, Multicenter Phase III Trial Evaluating the Efficacy and Safety of BCI-ImmuneActivator Versus Adriamycin in BCG Refractory or Intolerant Patients With Carcinoma in Situ With or Without Resected Superficial Papillary Bladder Cancer
Brief Title: Keyhole Limpet Hemocyanin Compared With Doxorubicin in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intracel (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: INTRACEL-BCI-9804-04; CDR0000068047 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-10-07 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2006-01

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — keyhole-limpet hemocyanin; Doxorubicin

ARMS (2):
- Arm I (Experimental): Patients receive a sensitizing dose of keyhole limpet hemocyanin (KLH) intradermally in week 2 followed by induction KLH IV once weekly in weeks 1-6. Patients with partial or no response receive IV KLH reinduction therapy once weekly in weeks 13-18. Patients with complete response receive IV KLH maintenance therapy monthly in weeks 13, 17, and 21, and then in months 6-12.
  Interventions: Biological: keyhole limpet hemocyanin
- Arm II (Active Comparator): Patients receive doxorubicin IV once weekly in weeks 1-6.
  Interventions: Drug: doxorubicin hydrochloride

INTERVENTIONS:
Biological: keyhole limpet hemocyanin — Given intradermally and IV
  Arms: Arm I
Drug: doxorubicin hydrochloride — Given IV
  Arms: Arm II

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether keyhole limpet hemocyanin is more effective than doxorubicin for bladder cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of keyhole limpet hemocyanin with that of doxorubicin in treating patients who have bladder cancer that has not responded to BCG or in those patients who cannot tolerate BCG.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of BCI-ImmuneActivator™ (keyhole limpet hemocyanin) versus doxorubicin in BCG refractory or intolerant patients with carcinoma in situ with or without resected superficial papillary bladder cancer.
* Compare the toxicity and safety of these treatments in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and prior BCG response (refractory vs intolerant). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive a sensitizing dose of keyhole limpet hemocyanin (KLH) intradermally at week -2 followed by induction KLH IV once weekly at weeks 1-6. Patients with partial or no response receive IV KLH reinduction therapy once weekly at weeks 13-18. Patients with complete response receive IV KLH maintenance therapy monthly at weeks 13, 17, and 21, and then at months 6-12.
* Arm II: Patients receive doxorubicin IV once weekly at weeks 1-6. Patients with complete response receive maintenance therapy comprising doxorubicin IV at weeks 13, 17, and 21 and months 6-12.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1.5 years, and then every 6 months for 1 year. (Patient total participation in this study may last as long as 42 months.)

PROJECTED ACCRUAL: A total of 150 patients (75 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed carcinoma in situ of the bladder with or without resected superficial papillary tumor

  * Biopsy within 3 months of study with or without positive urinary cytology within 6 weeks of study
* Cystoscopy within 3 months of study
* Negative imaging study of the ureters and kidneys within 6 months of study
* BCG refractory disease

  * Received and failed at least 1 prior induction course consisting of BCG weekly for 6 weeks OR
* BCG intolerant

  * Unable to receive an adequate course of intravesical BCG due to extreme toxicity
* Opted against or medically contraindicated to cystectomy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 11 g/dL

Hepatic

* Bilirubin normal
* SGOT/SGPT normal

Renal

* Creatinine no greater than 1.5 times upper limit of normal

Cardiovascular

* No severe cardiovascular disease

Other

* No other severe disease
* No other malignancy within the past 5 years except basal or squamous cell skin cancer or noninvasive cancer of the cervix
* No evidence of autoimmune disease, known immune deficiency, or immunosuppression
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior keyhole limpet hemocyanin immune activator

Chemotherapy

* No prior doxorubicin
* At least 3 months since prior mitomycin
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent steroids

Radiotherapy

* At least 4 months since prior radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 4 weeks since prior intravesical therapy
* At least 3 months since prior investigational agents
* No concurrent cytotoxic immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Hanna Jr., PhD, Study Chair — Intracel
Locations (1):
- Intracel Resources, LLC, Frederick, Maryland, United States